CLINICAL TRIAL: NCT03510520
Title: A Randomised Study Investigating the Effect of Medium Cut-Off Haemodialysis On Markers of Vascular Health Compared With On-Line HDF
Brief Title: Comparison of MCO HD on Markers of Vascular Health Compared With On-Line Haemodiafiltration
Acronym: MoDal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Manchester Metropolitan University (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R04863
Record Dates: First submitted 2018-04-12; First posted 2018-04-27 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: End Stage Renal Disease; Cardiovascular Diseases; Inflammation
Keywords: Hemodialysis; Haemodialysis; Hemodiafiltration; Haemodiafiltration; Dialysis membrane; Endothelial Microvesicles; Pulse Wave Velocity
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: This is a single-centre, pilot, open-label, interventional, randomised controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium Cut-Off Haemodialysis (Theranova) (Experimental): Participants will receive medium cut-off haemodialysis treatment for 6 months in total (3 times per week treatment).
  Interventions: Device: Medium Cut-Off Haemodialysis
- On-Line Haemodiafiltration (Active Comparator): Participant will remain on their usual on-line haemodiafiltration (HDF) treatment for the 6 month study duration (3 times per week treatment).
  Interventions: Device: On-Line Haemodiafiltration

INTERVENTIONS:
Device: Medium Cut-Off Haemodialysis — Treatment with medium cut-off haemodialysis using the Theranova dialysis membrane 3 times per week for 6 months
  Arms: Medium Cut-Off Haemodialysis (Theranova)
Device: On-Line Haemodiafiltration — Treatment with on-line haemodiafiltration (HDF) 3 times per week for 6 months (Conventional treatment)
  Arms: On-Line Haemodiafiltration

SUMMARY:
The aim of this study is to evaluate haemodialysis treatment using a medium cut-off dialysis membrane (Theranova) compared with on-line haemodiafiltration treatment with respect to markers of endothelial health (plasma endothelial microvesicle levels, pro-inflammatory and pro-coagulant markers).

This study will also compare the 2 treatment modalities with respect to several other outcome measures including patient-reported outcome measures, haemodynamic parameters and advanced glycation end-products.

DETAILED DESCRIPTION:
To date, methods of improving outcomes for haemodialysis patients have focused on improving small molecule clearance (urea); however, the benefits do not appear to be linear and increasing Kt/V above 1.3 shows no benefit. Current dialysis therapies are unable to provide effective clearance of larger "middle molecules" (between 20kDa and 60kDa) and retention of these molecules may be linked to poor outcomes in haemodialysis patients.

Medium cut-off (MCO) dialysis membranes have been recently developed to address this area of unmet need and provide an enhanced clearance of some larger middle molecules when compared with high flux haemodialysis (HFHD) and even high volume haemodiafiltration (HDF). The clinical benefit of this therapy is yet to be defined.

The aim of this study is to investigate the effect of HDx therapy (expanded haemodialysis therapy through the use of a MCO haemodialysis membrane- Theranova) on vascular endothelial and inflammatory biomarkers compared with high volume HDF therapy. Through the use of endothelial microvesicles (EMV) as a marker of vascular endothelial health, which strongly correlate with cardiovascular outcomes in end-stage real disease (ESRD) patients, this pilot study will take the first steps into exploring whether HDx treatment provides clinical benefits in addition to its simplicity of implementation. Additionally, other important parameters, such as dialysis recovery time, patient-reported outcome measures and volume management will also be explored and compared with high volume HDF.

ELIGIBILITY:
Inclusion Criteria:

* Established on in-centre haemodiafiltration (HDF) for greater than 12 weeks with a minimum of 3 treatment sessions per week
* Ability to consent

Exclusion Criteria:

* Planned live donor renal transplant within 6 months (with confirmed date)
* Planned switch in renal replacement modality (ie. to peritoneal dialysis or home haemodialysis)
* Clinician predicted prognosis < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function (composite of endothelial microvesicle levels, pro-inflammatory & pro-coagulant markers) | 6 months
  Change in vascular endothelial marker score (derived from multiple biomarkers)

SECONDARY OUTCOMES:
Change in pulse wave velocity | 6 months
  Change in pulse wave velocity as measured by non-invasive pulse wave analysis device
Change in pre-dialysis serum albumin | 3 & 6 months
  Change in pre-dialysis serum albumin
Change in pre-dialysis CRP | 3 & 6 months
  Change in pre-dialysis CRP
Change in components of pre-dialysis "middle molecule" panel | 3 & 6 months
  Change in components of pre-dialysis "middle molecule" panel (this includes beta 2 microglobulin, serum free light chains, leptin, beta trace protein and prolactin)
Change in components of cytokine panel | 3 & 6 months
  Change in components of cytokine panel (including IL-6, TNFa, ICAM & VEGF)
Change in numbers blood pressure medications | 6 months
  Change in numbers blood pressure medications
Change in number of phosphate binder medications | 6 months
  Change in number of phosphate binder medications
Change in Advanced Glycation End Products (AGE) | 6 months
  Change in Advanced Glycation End Products (AGE)
Change in inter-dialytic urine volume | 6 months
  Change in inter-dialytic urine volume
Change in IPOS-Renal (Integrated Palliative Care Outcome Score) | 3 & 6 months
  Change in IPOS-Renal (Integrated Palliative Care Outcome Score)
Change in self-sported dialysis recovery time | 3 & 6 months
  Change in self-sported dialysis recovery time
Change in Chalder fatigue scale | 3 & 6 months
  Change in Chalder fatigue scale (score range 0 to 33, high score indicating high levels of fatigue)
Hospitalisation episodes | 6 months
  Number of hospitalisation episodes during 6 months study period
All-cause mortality | 6 months
  All-cause mortality
Cardiovascular mortality | 6 months
  Cardiovascular mortality
Change in augmentation pressure (AP) | 6 months
  Change in segmentation pressure as measured by non-invasive pulse wave analysis device
Change in heart-rate adjusted augmentation index (AI) | 6 months
  Change in heart-rate adjusted augmentation index (AI) as measured by non-invasive pulse wave analysis device

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Mitra, MBBS, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester NHS Foundation Trust, Manchester, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is yet to be determined